CLINICAL TRIAL: NCT00003555
Title: Use of Weekly One Hour Paclitaxel Infusion With Dose Escalation for Recurrent and Resistant Cancers, Using Amifostine as a Cytoprotector
Brief Title: Paclitaxel Plus Chemoprotection With Amifostine in Treating Patients With Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: SUNY-HSC-3732; CDR0000066614 (Registry Identifier: PDQ (Physician Data Query)); ALZA-98-012-ii; NCI-V98-1463
Record Dates: First submitted 1999-11-01; First posted 2004-08-16 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2006-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Amifostine; Paclitaxel

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs, such as amifostine, may protect normal cells from the side effects of chemotherapy.

PURPOSE: Phase I trial to study the effectiveness of paclitaxel plus chemoprotection with amifostine in treating patients with recurrent or refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of weekly paclitaxel following amifostine in patients with recurrent or refractory solid tumors. II. Assess tumor response rate and survival in these patients.

OUTLINE: This is a dose escalation study of paclitaxel. Patients receive amifostine IV over 5 minutes or less on day 0, followed by paclitaxel IV over 1 hour once a week for 6 weeks followed by 2 weeks of rest. Patients with complete or partial response may receive additional courses of therapy. Cohorts of 3-5 patients each receive increasing doses of paclitaxel. The maximum tolerated dose is defined as the dose level prior to the cohort at which 1 of 3-5 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: Approximately 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent or refractory solid tumors Evaluable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Greater than 4 months Hematopoietic: Neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 8 g/dL Hepatic: Bilirubin less than 1.5 g/dL Alkaline phosphatase less than 3 times upper limit of normal (ULN) AST less than 3 times ULN Renal: Calcium greater than 8 mg/dL Creatinine clearance greater than 60 mL/min Cardiovascular: No active congestive heart failure Other: Not pregnant or nursing Fertile patients must use effective contraception No grade 2 neuropathy No intolerability for hydration

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior biologic therapy allowed Chemotherapy: No more than 3 prior failed chemotherapy regimens Prior paclitaxel as a radiosensitizer allowed No prior weekly paclitaxel infusion failure Prior platinum or paclitaxel therapy allowed Endocrine therapy: Prior endocrine therapy allowed Radiotherapy: Prior radiotherapy allowed Surgery: Prior surgery allowed Other: No concurrent dilantin therapy No antihypertensive/diuretics within 24 hours prior to chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1998-07; Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Wright, MD, Study Chair — State University of New York - Upstate Medical University
Locations (1):
- State University of New York - Upstate Medical University, Syracuse, New York, United States